CLINICAL TRIAL: NCT03248141
Title: UNDERSTANDING HEMOPHILIA A AND B DRUG DOSAGE ADMINISTRATION PATTERNS
Status: Terminated | Type: Observational
Why Stopped: Study recruitment was stopped due to difficulty in enrolling the targeted number of patients on March 21, 2018. See details in Description section.
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: B1821056; HEMOBAFS (Other: Alias Study Number)
Record Dates: First submitted 2017-05-31; First posted 2017-08-14 (Actual); Results first posted 2019-05-20 (Actual); Last update posted 2019-05-20 (Actual); Status verified 2019-02

CONDITIONS: Hemophilia A; Hemophilia B
Keywords: Hemophilia A Factor VIII; Hemophilia B Factor IX; Cross-sectional; Epidemiological; Clinical practice; United States
MeSH Terms: conditions — Hemophilia A; Hemophilia B

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Hemophilia B: real world administration patterns and resource utilization implications
  Interventions: Drug: Hemophilia B standard half-life; Drug: Hemophilia B extended half-life
- Hemophilia A: real world administration patterns and resource utilization implications
  Interventions: Drug: Hemophilia A standard half-life; Drug: Hemophilia A extended half-life

INTERVENTIONS:
Drug: Hemophilia B standard half-life — Benefix
  Groups: Hemophilia B
Drug: Hemophilia B extended half-life — Alprolix
  Groups: Hemophilia B
Drug: Hemophilia A standard half-life — Xyntha and other standard half-life agents
  Groups: Hemophilia A
Drug: Hemophilia A extended half-life — Eloctate and Adynovate
  Groups: Hemophilia A

SUMMARY:
Study Design

A prospective observational, cross-sectional epidemiological study in U.S. site-based clinical practice settings.

30 sites will enroll approximately 300 patients

Participating patients - or their caregiver in the case of patients under the age of 18 - will be consented to participate.

Physicians complete a retrospective chart review on each enrolled patient.

Patients will complete a one-time study questionnaire.

DETAILED DESCRIPTION:
Study recruitment was stopped due to difficulty in enrolling the targeted number of patients on March 21, 2018. Subjects currently enrolled into the study have completed the study as per protocol. There were no safety concerns involved in the decision to stop enrollment.

ELIGIBILITY:
Physician/Clinician Participants:

* Must be a healthcare provider
* Currently manages at least 10 hemophilia A and/or B patients

Patient Participants:

* Willing and able to provide informed consent
* Diagnosed with hemophilia A or B
* Current disease severity is either moderately severe or severe with a clotting factor level of ≤5%
* If suffering from hemophilia A, must be currently taking moroctocog alfa (or another standard half-life treatment), rurioctocog alfa or efraloctocog alfa for at least six months.

(If currently taking rurioctocog alfa or efraloctocog alfa, must have been switched from a standard half-life treatment and had been on that prior treatment for at least six months).

* If suffering from hemophilia B, must be currently taking nonacog alfa or eftrenonacog alfa for at least six months (If currently taking eftrenonacog alfa, must have switched from nonacog alfa and had been on that prior treatment for at least six months).
* Infuse at least 3 times per month

Exclusion criteria:

* Female with hemophilia A or B
* Mild Haemophilia A or B

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients diagnosed with either hemophilia A or B who present for a routine Clinical visit will be asked to participate in the study by the treating physician at participating hemophilia treatment centers in the United States of America.
Sampling Method: Non-Probability Sample
Enrollment: 11 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2018-03-14 (Actual); Study Completion 2018-03-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (3):
- United States (3):
  - University of Florida College of Medicine, Gainesville, Florida
  - Alliance for Childhood Diseases, dba Hemophilia Treatment Center of Nevada, Las Vegas, Nevada
  - Cook Children's Medical Center, Fort Worth, Texas

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B1821056&StudyName=Understanding+Hemophilia+A+And+B+Drug+Dosage+Administration+Patterns

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Out of 41 screened participants, 11 were enrolled in this study. Study got terminated afterwards due to difficulty in enrolling the targeted number of participants.
Groups:
- Hemophilia A Cohort: Participants diagnosed with Hemophilia A (disease severity either moderate: clotting factor level of less than and equal to [<=]5 percent[%] or severe: clotting factor level of less than [<]1%), and taking Xyntha or another standard half-life treatment (Adynovate or Eloctate) for at least 6 months (if taking Adynovate or Eloctate, must have been switched from a standard half-life treatment and had been on that prior treatment for at least six months and must have infused at least 3 times per month) were observed in this study for up to 6 months.
- Hemophilia B Cohort: Participants diagnosed with Hemophilia B (disease severity either moderate: clotting factor level <=5% or severe: clotting factor level of <1%), and taking BeneFIX or Alprolix for at least 6 months (if received Alprolix, must had switched from BeneFIX and had been on that prior treatment for at least 6 months and must have infused at least 3 times per month), were observed in this study for up to 6 months.
Period: Overall Study
Arm/Group | Hemophilia A Cohort | Hemophilia B Cohort
Started | 11 | 0 (No enrollment occurred in this arm prior to study termination.)
Completed | 11 (Participants who were present in the study till termination were considered as completed.) | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Analysis population included all enrolled participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Hemophilia A Cohort | Hemophilia B Cohort | Total
Number analyzed (Participants) | 11 | 0 | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 2 | 0 | 2
  Between 18 and 65 years | 9 | 0 | 9
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 11 | 0 | 11
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Resource Utilization Pattern
Time Frame: From baseline up to end of study (6 months)
Population: Data was not collected and analyzed for this outcome measure since very less number of participants were enrolled prior to study termination.
Arm/Group | Hemophilia A Cohort | Hemophilia B Cohort
Number analyzed (Participants) | 0 | 0

2. Primary Outcome: Dosing Pattern
Time Frame: From baseline up to end of study (6 months)
Population: as for outcome 1
Arm/Group | Hemophilia A Cohort | Hemophilia B Cohort
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: From baseline up to 6 months
Description: No enrollment occurred in Hemophilia B Cohort prior to study termination.
Arm/Group | Hemophilia A Cohort | Hemophilia B Cohort
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/0
Other Adverse Events (participants affected / at risk) | 0/11 | 0/0

LIMITATIONS AND CAVEATS:
Since study terminated early due to difficulty in enrolling targeted number of participants, so data was not collected and analyzed for any secondary endpoints, hence not reported in results. No safety concerns involved in decision to stop enrollment

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2017-04-04): https://cdn.clinicaltrials.gov/large-docs/41/NCT03248141/Prot_000.pdf
  • Statistical Analysis Plan (2017-04-17): https://cdn.clinicaltrials.gov/large-docs/41/NCT03248141/SAP_001.pdf